CLINICAL TRIAL: NCT04689438
Title: Usak University Faculty of Dentistry
Brief Title: GCF Levels of IL-1β and IL-6 in Gingivitis and Stage III-Grade C Periodontitis
Status: Completed | Type: Observational
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Ahu Dikilitaş, Usak University Faculty of Dentistry, Uşak University
Other Study IDs: UsakU7
Record Dates: First submitted 2020-12-28; First posted 2020-12-30 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Periodontitis
Keywords: periodontal disease; periodontitis; gingivitis; cytokines
MeSH Terms: conditions — Periodontitis; Periodontal Diseases; Gingivitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Gingival crevicular fluid
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy control groups: clinically healthy gingiva BOP score less than 10%
  Interventions: Diagnostic Test: gingival crevicular fluid
- Gingivitis groups: BOP score of 10% or greater
  Interventions: Diagnostic Test: gingival crevicular fluid
- Periodontitis groups: interdental AL ≥5 mm, PD≥6 mm
  Interventions: Diagnostic Test: gingival crevicular fluid

INTERVENTIONS:
Diagnostic Test: gingival crevicular fluid — GCF samples were collected in the morning hours 24-48 hours after clinical periodontal measurement.

SUMMARY:
Periodontal diseases are chronic diseases that occur as a result of a violation of the balance between microbial dental plaque and the host response. Gingivitis is a disease characterized by inflammation of the gingiva that occurs in one or more areas without loss of attachments.1 in periodontitis, an inflammatory event that begins in the gingiva along with gingivitis spreads to the periodontal ligament, alveolar bone and soft tissues that support the tooth, causing the destruction of these structures.2 Cytokines are low molecular weight proteins that participate in the initial and active stages of inflammation and immunity. In periodontal disease pathogenesis, cytokine response has been reported to play a very critical role in determining disease progression.3 IL-1beta and IL-6 are key cytokines in chronic inflammatory diseases and have the potential to initiate bone loss and tissue destruction seen in periodontal disease.4the purpose of this study; it is to determine the degree of inflammation and periodontal destruction by determining the levels of IL-1beta and IL-6 cytokines in the gingival crevicular fluid of periodontal healthy and diseased individuals.

DETAILED DESCRIPTION:
Periodontal measurement were done at 6 sites per tooth After clinical evaluation, individuals were divided into 3 groups

1. Healthy control groups:

   clinically healthy gingiva
2. Gingivitis groups:

   BOP score of 10% or greater and PD≤3mm
3. Periodontitis groups:

AL ≥5 mm, PD≥6 mm and tooth loss due to periodontitis of ≤4. GCF samples were collected using strips.

ELIGIBILITY:
Inclusion Criteria:

* have periodontitis
* have 16 permanent teeth

Exclusion Criteria:

* Systemic disease
* using drugs

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: individuals who have periodontal disease will be selected
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2020-12-25 (Actual); Study Completion 2020-12-28 (Actual)

PRIMARY OUTCOMES:
Measurement of IL-1Beta level | GCF was taken within 1 week after clinical examination
  GCF was taken interproximal region.
Measurement of IL-6 level in GCF | GCF was taken within 1 week after clinical examination
  GCF was taken interproximal region.

CONTACTS AND LOCATIONS:
Overall Officials: ahu dikilitaş, Principal Investigator — University of Usak; fatih karaaslan, Study Chair — University of Usak; abdullah seçkin ertuğrul, Study Chair — University of IZMIR KATİP CELEBİ
Locations (1):
- University of Usak, Uşak, Turkey (Türkiye)